CLINICAL TRIAL: NCT00836992
Title: Assessing the Clinical Significance of Real-time Quality of Life Data in Cancer Patients Treated With Radiation Therapy
Brief Title: Quality of Life in Patients Undergoing Radiation Therapy for Primary Lung Cancer, Head and Neck Cancer, or Gastrointestinal Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-005566; P30CA015083 (NIH); CDR0000629594 (Registry Identifier: NCI); 08-005566 (Other: Mayo Clinic IRB); MCS1065 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Anal Cancer; Colorectal Cancer; Esophageal Cancer; Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Head and Neck Cancer; Liver Cancer; Lung Cancer; Pancreatic Cancer; Small Intestine Cancer
Keywords: anal cancer; colon cancer; rectal cancer; esophageal cancer; extrahepatic bile duct cancer; gallbladder cancer; gastric cancer; adult primary liver cancer; pancreatic cancer; small intestine cancer; non-small cell lung cancer; small cell lung cancer; head and neck cancer
MeSH Terms: conditions — Anus Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Patient's QOL assessments data is not shared with the physician, nurse, and/or nurse practitioner and the patient
- Active: Patient's QOL assessments data is shared with the physician, nurse, and/or nurse practitioner and the patient immediately prior to the on-treatment visit.

SUMMARY:
RATIONALE: Gathering information about patients' quality of life during radiation therapy for cancer may help doctors plan the best treatment.

PURPOSE: This randomized clinical trial is studying quality of life in patients undergoing radiation therapy for primary lung cancer, head and neck cancer, or gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if patient-reported quality of life (QOL) can be improved by the real-time use of QOL data in patients with primary lung, head and neck, or gastrointestinal cancer undergoing radiotherapy.
* To obtain preliminary estimates for effect sizes on differences in key QOL domains between patients receiving real time QOL data and those not receiving QOL data.
* To obtain preliminary estimates of differences in patient satisfaction between patients receiving real time QOL data and those not receiving QOL data.
* To determine whether the availability of real-time QOL assessments in a radiation oncology practice increases the acceptance and utilization of QOL data by a clinical oncology team.
* To evaluate clinician attitudes towards the incorporation of real-time QOL data into oncology patient management.
* To evaluate the use of a set of clinical pathways for the incorporation of real time QOL data into oncology patient management.
* To evaluate the potential impact on the quality of the patient-physician relationship with real-time use of QOL data compared to interactions where quality of life data are not utilized.
* To obtain preliminary estimates of whether the real-time use of QOL data in a radiation oncology practice significantly increases the duration of the weekly on treatment visit.

OUTLINE: Patients are randomized to 1 of 2 groups.

* Group 1 (control): Patients complete QOL assessments (e.g., the Linear Analog Self Assessment [LASA]) at weeks 1, 3, and 5 during treatment and the last week of treatment. They also complete the Interpersonal Patient-Provider Relationship Scale (IPPRS) and Was it Worth It (WIW) questionnaires on the final day of treatment. Data is not shared with the physician, the patient, or any other clinical assistant that may be supporting the physician (e.g. nurse, or nurse practitioner).
* Group 2 (active): Patients complete QOL assessments (e.g., LASA) and the IPPRS and WIW questionnaires as in group 1. Information from the questionnaires is shared with the physician, nurse, and/or nurse practitioner and the patient immediately prior to the on-treatment visit.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Primary lung cancer
  * Head and neck cancer
  * Gastrointestinal cancer
* No evidence of distant metastasis
* Receiving ≥ 5 weeks of definitive or adjuvant radiotherapy at Mayo Clinic Arizona

PATIENT CHARACTERISTICS:

* Able to complete computer based questionnaires
* Able to complete quality of life questionnaires in English
* Willing and able to comprehend and provide informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck tumors, lung tumors, and gastrointestinal tumors receiving radiation therapy at Mayo Clinic Arizona
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2011-09-15 (Actual); Study Completion 2015-07-27 (Actual)

PRIMARY OUTCOMES:
Overall quality of life (QOL) scores at baseline, weeks 1, 3, 5, and end of treatment as assessed by LASA | 7 Weeks

SECONDARY OUTCOMES:
Component QOL domains reported on the five numerical analogue items (physical, intellectual, emotional, spiritual, and social QOL), average pain item and fatigue reported in the LASA | 7 Weeks
Frequency and severity of toxicity as assessed by NCI CTCAE at baseline, weeks 1, 3, 5, and of treatment | 7 Weeks
Scores from the IPPRS, satisfaction with the physician scale score, and global question assessment | 7 Weeks
Quantitative assessments from the post-treatment questionnaires and the qualitative data gleaned from the post-treatment interviews | One month post study
Proportion of cases for which the clinical team indicates that the clinical pathways contributed positively to patient management, the number of cases which the clinicians report referrals were generated, and the qualitative data derived from the pos ... | One month post study
Average physician rating of the patient-physician relationships for the two treatment groups | 7 Weeks
Average duration of the weekly on treatment visit for the two treatment groups | 7 Weeks
Percentage of patients for which physician reports indicate that availability | 7 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michele Yvette Halyard, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States